CLINICAL TRIAL: NCT03244150
Title: Youth and Sport Study - a 20 Year Follow-up Study of Danish Teenagers Born Between 1964 and 1969
Brief Title: Youth and Sport Study
Acronym: YSS
Status: Completed | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Collaborators: the Danish Medical Research Council (grant number 09-060078/FSS) (Unknown); The Danish Ministry of Health (2003-0200-13) (Unknown); Aase and Ejnar Danielsens Foundation (Other); The Copenhagen Hospital Corporation (now Copenhagen Capital Region) (Unknown)
Responsible Party: Principal Investigator, Berit Lilienthal Heitmann, Professor, Ph.D, Bispebjerg Hospital
Other Study IDs: 09-060078/FSS; 2003-0200-13 (Other Grant/Funding Number: The Danish Ministry of Health)
Record Dates: First submitted 2017-07-31; First posted 2017-08-09 (Actual); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Physical Activity; Obesity; Lifestyle
Keywords: Physical activity; Obesity; Overweight; Lifestyle; Diet
MeSH Terms: conditions — Motor Activity; Obesity; Overweight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA samples were collected by cheek scrapings, which were distributed and returned through mail.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- School sample: Conducted in 1983 and included 1260 students in high school or trade school.
- Nationwide sample: Conducted in 1985 and included a representative sample of 2498 teenagers drawn from the Danish Civil Registration (CPR)

SUMMARY:
The Youth and Sport Study (YSS) is a 20-22-year follow-up study of Danish teenagers born between 1964 and 1969. Baseline data originate from two different studies carried out in 1983 and 1985, and the follow-up study was carried out in 2005.

DETAILED DESCRIPTION:
The first baseline study was conducted in 1983 and included 1260 students in high school or trade school. The questionnaire was designed with focus on various aspects of sports and physical activity beside more general questions on family, socioeconomic status, height, weight, alcohol intake, smoking, etc. Furthermore, the participants were subjected to a set of physical tests and measurements.

The second baseline study was conducted in 1985 and included a representative sample of 2498 teenagers drawn from the Danish Civil Registration (CPR) and invited to participate in the study with the aim of validating the results from the first baseline sample. The study consisted of a questionnaire with virtually the same questions as the questionnaire from 1983. A short 28-item food frequency questionnaire (FFQ) was added to the questionnaire, as well as a few questions about dietary habits.

The follow-up study was carried out in 2005, when the subjects had reached an age of around 40 years. A total of 1904 subjects were traced and asked to complete a general questionnaire, a food frequency questionnaire, and deliver a DNA sample, all distributed and returned through mail correspondence. The general questionnaire included questions on education, occupation, height, previous and present weight, weight loss history, physical activity, smoking, civil status, children, other family, stress, diseases, hospital admissions, and medicine use, among other things. The questions about physical activity were adopted from the baseline questionnaire. Other questions were adopted from other validated questionnaires. Moreover, a semi-quantitative, 195-item Food Frequency Questionnaire (FFQ), which previously has been used and validated in the Danish "Diet, Cancer and Health" study was included. The study was approved by the local ethics committee for Copenhagen and Frederiksberg (J.nr. KF 01-260/04).

ELIGIBILITY:
Danish teenagers born between 1964 and 1969.

Ages: 15 Years to 19 Years | Sex: All
Age Groups: Child, Adult
Study Population: The first baseline study included 1260 students in gymnasium, vocational school, or trade school born in 1964-68.
  The second baseline study included a representative sample of 2498 teenagers born in 1967 or 1969 (1.5% of the total population).
Sampling Method: Probability Sample
Enrollment: 3008 (Actual)
Dates: Start 1983-08-01 (Actual); Primary Completion 2005-08-01 (Actual); Study Completion 2005-08-01 (Actual)

PRIMARY OUTCOMES:
Physical activity | Collected/measured in 1983 or 1985 and at follow-up in 2005
  Leisure time physical activity has been assessed by questionnaire, where participants filled in the different types of sports they attended and the time they actively participated in each type of sport per week. Lastly, the type and the amount of time spend on activities outside of school and sports clubs were also assessed. Each sport and activity has been translated into metabolic equivalent (MET) scores [28]. MET scores at the individual time points and changes during follow-up will be used as outcome.

SECONDARY OUTCOMES:
Body Mass Index (BMI) | Weight was reported in 1983 or 1985 and at follow-up in 2005
  BMI will be calculated using self-reported height and weight for both baseline and follow-up surveys. BMI at the individual time points and changes during follow-up will be used as outcome.
Waist circumference | Waist circumference was at follow-up in 2005
  Waist circumference was self-reported at the follow-up survey.
Alcohol consumption | Alcohol consumption was reported in 1983 or 1985 and at follow-up in 2005
  Alcohol consumption was assessed by the question "How often do you drink different types of alcohol?" with three choices - beer, wine and spirit". Alcohol at the individual time points and changes during follow-up will be used as outcome.
Smoking | Information on smoking was reported in 1983 or 1985 and at follow-up in 2005
  Smoking was assessed with the questions on smoking status and amount of tobacco smoked at baseline and follow-up. Information on smoking at the individual time points and changes during follow-up will be used as outcome.
Education and occupation | Information on education and occupation was reported in 2005
  At follow-up, participants were asked to report their occupation and highest achieved education.
Parental education and occupation | Information on education and occupation was reported in 1983 or 1985
  At baseline, participants were asked to report parental occupation and highest education.
Macronutrient intake | Information on macronutrient intake was reported in 2005
  At follow-up, participants completed a 28-item food frequency questionnaire. From this we will calculate the participants' macronutrient intake.

CONTACTS AND LOCATIONS:
Locations (1):
- Parker Institute, Frederiksberg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Poudel P, Ismailova K, Andersen LB, Larsen SC, Heitmann BL. Adolescent wine consumption is inversely associated with long-term weight gain: results from follow-up of 20 or 22 years. Nutr J. 2019 Sep 10;18(1):56. doi: 10.1186/s12937-019-0478-7. PMID 31506084